CLINICAL TRIAL: NCT03841539
Title: Enhanced Mediterranean Diet for Alzheimer's Disease Prevention
Brief Title: Nutrition Interventions for Cognitive Enhancement
Acronym: NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Debra K. Sullivan, PhD, RD, Chair and Endowed Professor of Clinical Nutrition, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00142752; 1R01AG060157-01 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-02-15 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
Keywords: Cognitive Impairment; Dementia; Alzheimer Disease; Mediterranean Diet; Low Fat Diet
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a dietary intervention; Mediterranean or Low-Fat, and will follow this eating pattern for 12 months.
Who Masked: Outcomes Assessor
Masking Description: Raters - (psychometrician, brain magnetic resonance imaging (MRI), dual energy x-ray absorptiometry (DEXA), and phlebotomy) will be blinded to the intervention group and will perform outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Experimental): Follow a Mediterranean eating pattern and take a study supplement for one year. Dietary education will be provided by a Registered Dietitian.
  Interventions: Behavioral: Mediterranean Diet; Dietary Supplement: Study Supplement
- Low-fat Diet (Active Comparator): Follow a low-fat eating pattern and take a study supplement for one year. Dietary education will be provided by a Registered Dietitian.
  Interventions: Dietary Supplement: Study Supplement; Behavioral: Low-fat Diet

INTERVENTIONS:
Behavioral: Mediterranean Diet — Diet consisting of fruits, vegetables, whole grains, low-fat dairy, olive oil, seafood, nuts and beans. It is low in red and processed meats, solid fats and added sugars.
  Arms: Mediterranean Diet
Dietary Supplement: Study Supplement — Randomized to take a daily dose of either 2 grams of Omega 3 fatty acids or 2 grams of a Placebo.
Behavioral: Low-fat Diet — Diet consisting of fruits, vegetables, whole grains, low-fat dairy, and low-fat protein, with fat contributing no more than 25% of calories.
  Arms: Low-fat Diet

SUMMARY:
By doing this study, researchers hope to learn how the Mediterranean and low-fat eating patterns affect memory, brain volume, brain antioxidant status and cardio-metabolic biomarkers, such as blood pressure and blood glucose, in cognitively normal older adults. Researchers also plan to examine underlying processes relating the patterns to brain health.

DETAILED DESCRIPTION:
Participants will be randomized to either a Mediterranean or low-fat eating pattern. Participation in the study will last about 13 months. Each person will be prescribed one of two eating patterns for 12 months. During the study, participants will be asked to track the food they eat and will be monitored by a registered dietitian. Participants will engage in monthly food demonstrations and cooking classes. Participants will pick up a bag of food items belonging to the prescribed eating pattern, on a weekly basis for 6 months, from a local grocery store chain.

Participants have the option to continue in the study for up to 2 years for additional measurements.

Potential participants need to be located within the Kansas City metro area.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal older adults ≥65 years (MMSE score ≥ 25; AD8 score of 2 or less; no prior diagnosis of MCI, AD or dementia; and not medically treated for cognitive impairment or dementia)
* Speak English as a primary language
* Be able to read and write in English
* Live in the Kansas City, Metropolitan area
* Body Mass Index (BMI) range between 20 - 40 kg/m2

Exclusion Criteria:

* Serious medical risk, such as type 1 diabetes mellitus, cancer, recent cardiac event (e.g. heart attach, angioplasty)
* Taking the prescription drug Warfarin
* Taking a prescription fish oil, such as Lovaza, Omtryga, Vascepa, Epanova, etc., or prescribed a dose of over-the-counter (OTC) fish oil containing ≥300 mg Docohexanoic Acid (DHA) that cannot be adjusted to a lower dose
* Nut allergy, fish allergy (does not include shellfish)
* Adherence to specialized diet regimes (e.g., vegan, bariatric, renal, etc.) that make following either of the dietary plans impossible or unsafe
* Unwilling to be randomized to one of two diet interventions
* Evidence of severe major depression (GDS-SF ≥9) or presence of a major psychiatric disorder that in the investigator's opinion, could interfere with adherence to research assessments or procedures
* Alcohol (over 3 drinks per day or total of 18 per week) or drug abuse, defined as the use of chemical substances (prescription, OTC or illegal drugs) in a pattern that can lead to an increased risk of problems and an inability to control the use of the substance
* Do not have access to or independence over grocery shopping and meal preparation (i.e. those in military, retirement community with reliance on dining facilities for meals)
* Already consuming a Mediterranean diet as determined using the 14-item MedD Assessment Tool (score of ≥8)
* Already consuming a low-fat diet as determined by the NCI Percentage Energy from Fat Screener (≤ 15% of calories from fat)
* Already participating in another research study
* Another member of household is already participating in this study
* Have a visual impairment that greatly diminishes ability to read or write
* Currently attempting to lose weight

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 209 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Change in a composite global cognition score | Baseline, 6 months and 12 months
  Alzheimer's Disease Cooperative Study-Preclinical Alzheimer Cognitive Composite (ADCS-PACC) and NIH Toolbox (NIH-TB) Cognition Battery and will be used to assess changes in a composite global cognition score at baseline, 6, and 12 months.

SECONDARY OUTCOMES:
Change in Verbal Memory Factor | Baseline, 6 months and 12 months
  Change in Verbal Memory Factor (derived from confirmatory factor analyses (CFA) of the following scales: Logical Memory I, Logical Memory II, and Selective Reminding Task) at baseline, 6 months and 12 months. CFA aggregates scores from across multiple subtests.
Change in Visuospatial Processing Factor | Baseline, 6 months and 12 months
  Change in Visuospatial Processing Factor (derived from confirmatory factor analyses (CFA) of the following scales: Stroop Color Naming, Digit Symbol, Block Design, and Trailmaking A) at baseline, 6 months and 12 months. CFA aggregates scores from across multiple subtests.
Change in Attention Factor | Baseline, 6 months and 12 months
  Change in Attention Factor (derived from confirmatory factor analyses (CFA) of the following scales: Digits Forward, Digits Backward, and Letter-Number Sequencing) at baseline, 6 months and 12 months. CFA aggregates scores from across multiple subtests.
Change in Executive Function Factor | Baseline, 6 months and 12 months
  Change in Executive Function Factor (derived from confirmatory factor analyses (CFA) of the following scales: NIH-TB Dimensional Change Card Sort Test, NIH-TB Flanker Inhibitory Control and Attention Test, Trailmaking B, and Category Fluency) at baseline, 6 months and 12 months. CFA aggregates scores from across multiple subtests.
Change in Speed of Processing Factor | Baseline, 6 months and 12 months
  Change in Speed of Processing Factor (derived from confirmatory factor analyses (CFA) of the following scales: of Crossing Off and NIH-TB Pattern Comparison Processing Speed Test) at baseline, 6 months and 12 months. CFA aggregates scores from across multiple subtests.
Change in brain volume | Baseline and 12 months
  Change in whole brain and hippocampal volume as assessed via magnetic resonance imaging (MRI) at baseline and 12 months.
Change in cerebral antioxidant levels | Baseline and 12 months
  Antioxidant levels are measured in frontal and parietal regions of the brain using magnetic resonance spectroscopy in a 3 T clinical scanner.
Change in blood pressure | Baseline, 6 months and 12 months
  Measure of both systolic blood pressure and diastolic blood pressure at baseline, 6 months, and 12 months.
Change in percentage of total fatty acids by weight | Baseline and 12 months
  Measure of red blood cell (RBC)-phospholipids at baseline and 12 months.
Change in total cholesterol | Baseline and 12 months
  Measure of total cholesterol at baseline and 12 months
Change in HDL cholesterol | Baseline and 12 months
  Measure of HDL cholesterol at baseline and 12 months
Change in total/HDL cholesterol ratio | Baseline and 12 months
  Measure of total/HDL cholesterol ratio at baseline and 12 months
Change in LDL cholesterol | Baseline and 12 months
  Measure of LDL cholesterol at baseline and 12 months
Change in triglycerides | Baseline and 12 months
  Measure of triglycerides at baseline and 12 months
Change in apolipoprotein B | Baseline and 12 months
  Measure of apolipoprotein B, a measure of cardiovascular disease risk, at baseline and 12 months
Change in lipoprotein(a) (Lp(a)) | Baseline and 12 months
  Measure of Lp(a), a measure of cardiovascular disease risk, at baseline and 12 months
Change in high sensitivity C-Reactive Protein (hs-CRP) | Baseline and 12 months
  Measure of hs-CRP, a measure of inflammation, at baseline and 12 months
Change in lipoprotein-associated phospholipase A2 (Lp-PLA2) | Baseline and 12 months
  Measure of Lp-PLA2 activity, a measure of cardiovascular disease risk, at baseline and 12 months
Change in insulin resistance score | Baseline and 12 months
  Measure of intact insulin and c-peptide to determine an insulin resistance score at baseline and 12 months
Change in fasting glucose | Baseline and 12 months
  Measure of glucose at baseline and 12 months
Change in Hemoglobin A1c (HbA1c) | Baseline and 12 months
  Measure of HbA1c at baseline and 12 months
Change in Trimethylamine N-oxide (TMAO) | Baseline and 12 months
  Measure of TMAO, a measure of cardiovascular disease risk, at baseline and 12 months
Change in a composite global cognition score post intervention | 24 and 36 months
  Alzheimer's Disease Cooperative Study-Preclinical Alzheimer Cognitive Composite (ADCS-PACC) and NIH Toolbox (NIH-TB) Cognition Battery and will be used to assess changes in a composite global cognition score at 24 and 36 months.
Change in Verbal Memory Factor post intervention | 24 and 36 months
  Change in Verbal Memory Factor (derived from confirmatory factor analyses (CFA) of the following scales: Logical Memory I, Logical Memory II, and Selective Reminding Task) at 24 and 36 months. CFA aggregates scores from across multiple subtests.
Change in Visuospatial Processing Factor post intervention | 24 and 36 months
  Change in Visuospatial Processing Factor (derived from confirmatory factor analyses (CFA) of the following scales: Stroop Color Naming, Digit Symbol, Block Design, and Trailmaking A) at 24 and 36 months. CFA aggregates scores from across multiple subtests.
Change in Attention Factor post intervention | 24 and 36 months
  Change in Attention Factor (derived from confirmatory factor analyses (CFA) of the following scales: Digits Forward, Digits Backward, and Letter-Number Sequencing) at 24 and 36 months. CFA aggregates scores from across multiple subtests.
Change in Executive Function Factor post intervention | 24 and 36 months
  Change in Executive Function Factor (derived from confirmatory factor analyses (CFA) of the following scales: NIH-TB Dimensional Change Card Sort Test, NIH-TB Flanker Inhibitory Control and Attention Test, Trailmaking B, and Category Fluency) at 24 and 36 months. CFA aggregates scores from across multiple subtests.
Change in Speed of Processing Factor post intervention | 24 and 36 months
  Change in Speed of Processing Factor (derived from confirmatory factor analyses (CFA) of the following scales: of Crossing Off and NIH-TB Pattern Comparison Processing Speed Test) at 24 and 36 months. CFA aggregates scores from across multiple subtests.
Measure of dietary adherence post intervention | 24 and 36 months
  Measure of dietary adherence through 3 day food records at 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Sullivan, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No